CLINICAL TRIAL: NCT04213716
Title: Comparison of the Efficacy of Calcium Hydroxide Combined With Silver Nano Particulate and Conventional Calcium Hydroxide Intra Canal Medications on Post-Operative Pain in Symptomatic Root Canal Treatment Failure Cases: A Randomized Clinical Trial Therapeutic Study
Brief Title: Comparison of the Efficacy of Calcium Hydroxide With Silver Nanoparticle and Conventional Calcium Hydroxide Intra Canal Medications on Post-Operative Pain in Symptomatic Root Canal Treatment Failure Cases:
Acronym: CSNIMSRRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawda Mohammad Abdel Rahman Baghdady, cairo egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO-CU-2014-9-14
Record Dates: First submitted 2019-12-21; First posted 2019-12-30 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Retreatment; Root Canal Retreatment; Nonsurgical Retreatment; Endodontic Failure; Symptomatic Endodontic Failure; Nanosilver; Intracanal Medicament; Intracanal Dressing; AgNPs; Calcium Hydroxide; Ca (OH)2; Discomfort; Pain; Flare up; Postoperative; Ache; Post-operative; Post Obturation
Keywords: Keywords provided by rawda mohammad abdel rahman baghdady, Cairo University:; root canal retreatment; calcium hydroxide; distilled water; silver nanoparticles; postoperative pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Interventions: (60) Intracanal medication of 1ml combined nanosilver particle solution 30ppm / 100 mg calcium hydroxide Control : (60) Intracanal medication of 100 mg powder of calcium hydroxide mixed with 1ml distilled water
Who Masked: Participant, Outcomes Assessor
Masking Description: Bottles of nanosilver solution & distalled water will be covered and coded either A or B by assistant supervisor, and then given to the operator.
  Participants will be blinded as regard to either intervention or control Participant and operator who is also the outcome assessor are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intracanal medication (Experimental): After instrumentation of the canals and drying , using Lentulo Spiral Filler medicaments will be placed under aseptic conditions into the canals experimental Intracanal medication of 1ml of nanosilver solution 30ppm concentration mixed with 100 mg of calcium hydroxide powder used as intracanal medication
  Interventions: Combination Product: silver nano particulate solution mixed with calcium hydroxide powder
- intracanal medicament (Active Comparator): After instrumentation of the canals and drying , using Lentulo Spiral Filler comparator intracanal medicaments will be placed under aseptic conditions into the canals which is 100 mg Ca (OH) 2 mixed with 1ml sterile water
  Interventions: Combination Product: conventional calcium hydroxide

INTERVENTIONS:
Combination Product: silver nano particulate solution mixed with calcium hydroxide powder — 1ml of nanosilver solution 30ppm concentration mixed with 100 mg of calcium hydroxide powder used as intracanal medication
  Arms: intracanal medication
Combination Product: conventional calcium hydroxide — 1ml of distilled water mixed with 100 mg of calcium hydroxide powder and used as intracanal medication after root canal retreatment
  Arms: intracanal medicament

SUMMARY:
The aim of this study is to measure and compare the effectiveness of nanosilver combined calcium hydroxide and conventional calcium hydroxide intracanal medications in reducing postoperative pain in patients with Symptomatic Root Canal treatment Failure .

DETAILED DESCRIPTION:
* After confirming the diagnosis and making sure that the patient conforms to all eligibility criteria, the principal investigator will enroll the patient in the study.
* The operator will complete treatment of all cases in two visits as follows:

  1. First session:

     * Patients will be asked to rate their pain level on NRS before treatment is started.
     * Patient will be anesthetized by using nerve block local anesthesia or infiltration local anesthesia according to the tooth location in mandibular or maxillary arch respectively.
     * Previous coronal restoration will be removed:

       * If the access will be cut through metal (amalgam alloy or cast metal) or composite resin, carbide fissure bur will be used.
       * In case of porcelain fused to metal (PFM) crown a round diamond is used to cut through the porcelain layer, then Transmetal bur is used to cut through and remove the core material.
     * Teeth will be isolated with rubber dam.
     * Gutta percha removal will be done using protaper rotary retreatment files in the following manner D1 has a cutting tip to facilitate initial penetration into the filling material (coronal third). D2 and D3 both have non-cutting tips and are used to remove material from the middle and apical thirds, respectively using gutta percha solvent
     * Working length will be determined using an electronic apex locator then confirmed with intraoral periapical radiograph, to be 0.5-1 mm, shorter than radiographic apex.
     * Cleaning and shaping will be done using crown down preparation technique with the use of protaper rotary files in an endodontic motor according to the manufacturer instructions, the canals will be thoroughly irrigated using 3ml of 2.5% Sodium hypochlorite between every subsequent instruments.
     * MD-Chelcream will be used as lubricant during mechanical preparation.
     * After instrumentation of the canals paper points (Protaper Paper Points) will be used for drying.
     * Using Lentulo Spiral Filler, medicaments will be placed under aseptic conditions into the canals according to each group, Experimental group Ca (OH) 2 ( Ca (OH) 2with nanosilver suspension and comparison group Ca (OH) 2 with sterile water then access cavity will be closed with a temporary filling
     * Patient will be instructed to call in case of severe pain in between visits, an emergency analgesics are to be prescribed to the patient (Brufen 400mg)
  2. Second session:

     * After 7 days, rubber dam will be placed , the temporary fillings will be removed and master apical file will be introduced in each root canal to loosen medicament and to create a space for subsequent irrigant, then each root canal will be washed with 5 mL of sterile saline, irrigated with 1 mL of 20% citric acid and again irrigated with 5 mL sterile saline.
     * Dryness of the canals by paper points (Protaper Paper Points).
     * Obturation will be carried out using the cold lateral condensation technique with protaper gutta percha cones and resin sealer with spreader size according to master cone size , its depth short 2 mm of the working length, and auxiliary cones size 25.
     * After obturation a cotton pellet will be placed in the pulp chamber and the access cavity will be closed with a temporary filling to avoid coronal leakage.
     * The patient is given a NRS and asked to rate his pain level at 6, 12, 24 & 48 hours after root canal retreatment .

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients.
* Patient's age between 25-50 years.
* Anterior or premolar teeth diagnosed clinically and radio graphically as symptomatic root canal treatment failure.
* Positive patient's acceptance for participation in the study.
* Sex include both male and female.
* Patients who can understand Numerical Rating Scale (NRS)
* Patients able to sign informed consent.

Exclusion Criteria:

* Pregnancy or lactation.
* Medically compromised patients.
* Patient with multiple teeth that required retreatment to eliminate the possibility of pain referral.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain using a pain-measuring scale | [ Time Frame:6 hours ]
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 6 hours after the second visit (after obturation)
Postoperative pain using a pain-measuring scale | [ Time Frame: 12 hours ]
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 12 hours after the second visit (after obturation)
Postoperative pain using a pain-measuring scale | [ Time Frame: 24 hours ]
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 24 hours after the second visit (after obturation)
Postoperative pain using a pain-measuring scale | [ Time Frame: 48 hours ]
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 48 hours after the second visit (after obturation)

CONTACTS AND LOCATIONS:
Overall Officials: Rawda baghdady, M.S.c, Principal Investigator — Cairo University; Jealan El shafei, professor, Study Director — Cairo University; Alaa El baz, assist prof, Study Chair — Cairo University
Locations (1):
- Endodontic Department , Faculty of Dentistry , Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siqueira JF Jr. Aetiology of root canal treatment failure: why well-treated teeth can fail. Int Endod J. 2001 Jan;34(1):1-10. doi: 10.1046/j.1365-2591.2001.00396.x. PMID 11307374
- [Background] Daokar DS, Kalekar DA "Endodontic Failures-A Review," Journal of Dental and Medical Sciences 4(5): 5-10, 2013
- [Background] Siqueira JF Jr, Rocas IN, Favieri A, Machado AG, Gahyva SM, Oliveira JC, Abad EC. Incidence of postoperative pain after intracanal procedures based on an antimicrobial strategy. J Endod. 2002 Jun;28(6):457-60. doi: 10.1097/00004770-200206000-00010. PMID 12067129
- [Background] Peciuliene V, Reynaud AH, Balciuniene I, Haapasalo M. Isolation of yeasts and enteric bacteria in root-filled teeth with chronic apical periodontitis. Int Endod J. 2001 Sep;34(6):429-34. doi: 10.1046/j.1365-2591.2001.00411.x. PMID 11556508
- [Background] Gama TG, de Oliveira JC, Abad EC, Rocas IN, Siqueira JF Jr. Postoperative pain following the use of two different intracanal medications. Clin Oral Investig. 2008 Dec;12(4):325-30. doi: 10.1007/s00784-008-0199-3. Epub 2008 Apr 10. PMID 18401602
- [Background] Singh RD, Khatter R, Bal RK, Bal CS. Intracanal medications versus placebo in reducing postoperative endodontic pain--a double-blind randomized clinical trial. Braz Dent J. 2013;24(1):25-9. doi: 10.1590/0103-6440201302039. PMID 23657409
- [Background] Kawashima N, Wadachi R, Suda H, Yeng T, Parashos P. Root canal medicaments. Int Dent J. 2009 Feb;59(1):5-11. PMID 19323305
- [Background] Wu D, Fan W, Kishen A, Gutmann JL, Fan B. Evaluation of the antibacterial efficacy of silver nanoparticles against Enterococcus faecalis biofilm. J Endod. 2014 Feb;40(2):285-90. doi: 10.1016/j.joen.2013.08.022. Epub 2013 Oct 1. PMID 24461420
- [Background] M. Mustafa, D. Jain, M. Kadri and etal. , " Role of Calcium Hydroxide in Endodontics : A Review," Global Journal of Medical and Public Health,vol. 1, no. 1, pp. 53-57, 2012.
- [Background] Silveira CF, Cunha RS, Fontana CE, de Martin AS, Gomes BP, Motta RH, da Silveira Bueno CE. Assessment of the antibacterial activity of calcium hydroxide combined with chlorhexidine paste and other intracanal medications against bacterial pathogens. Eur J Dent. 2011 Jan;5(1):1-7. PMID 21311611
- [Background] Pacios MG, Silva C, Lopez ME, Cecilia M. Antibacterial action of calcium hydroxide vehicles and calcium hydroxide pastes. J Investig Clin Dent. 2012 Nov;3(4):264-70. doi: 10.1111/j.2041-1626.2012.00147.x. PMID 23129141
- [Background] Vianna ME, Gomes BP, Sena NT, Zaia AA, Ferraz CC, de Souza Filho FJ. In vitro evaluation of the susceptibility of endodontic pathogens to calcium hydroxide combined with different vehicles. Braz Dent J. 2005;16(3):175-80. doi: 10.1590/s0103-64402005000300001. Epub 2006 Jan 12. PMID 16429180
- [Background] Yoldas O, Topuz A, Isci AS, Oztunc H. Postoperative pain after endodontic retreatment: single- versus two-visit treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Oct;98(4):483-7. doi: 10.1016/j.tripleo.2004.03.009. PMID 15472665
- [Background] Adl A, Hamedi S, Sedigh Shams M, Motamedifar M, Sobhnamayan F. The ability of triple antibiotic paste and calcium hydroxide in disinfection of dentinal tubules. Iran Endod J. 2014 Spring;9(2):123-6. Epub 2014 Mar 8. PMID 24688581
- [Background] Cwikla SJ, Belanger M, Giguere S, Progulske-Fox A, Vertucci FJ. Dentinal tubule disinfection using three calcium hydroxide formulations. J Endod. 2005 Jan;31(1):50-2. doi: 10.1097/01.don.0000134291.03828.d1. PMID 15614007
- [Background] Javidi M, Afkhami F, Zarei M, Ghazvini K, Rajabi O. Efficacy of a combined nanoparticulate/calcium hydroxide root canal medication on elimination of Enterococcus faecalis. Aust Endod J. 2014 Aug;40(2):61-5. doi: 10.1111/aej.12028. Epub 2013 May 12. PMID 25244219
- [Background] Mei L, Lu Z, Zhang W, Wu Z, Zhang X, Wang Y, Luo Y, Li C, Jia Y. Bioconjugated nanoparticles for attachment and penetration into pathogenic bacteria. Biomaterials. 2013 Dec;34(38):10328-37. doi: 10.1016/j.biomaterials.2013.09.045. Epub 2013 Sep 30. PMID 24090838
- [Background] Mohammadi Z, Soltani MK, Shalavi S. An update on the management of endodontic biofilms using root canal irrigants and medicaments. Iran Endod J. 2014 Spring;9(2):89-97. Epub 2014 Mar 8. PMID 24688576
- [Background] Imura N, Zuolo ML. Factors associated with endodontic flare-ups: a prospective study. Int Endod J. 1995 Sep;28(5):261-5. doi: 10.1111/j.1365-2591.1995.tb00311.x. PMID 8626209
- [Background] Seltzer S, Naidorf IJ. Flare-ups in endodontics: I. Etiological factors. 1985. J Endod. 2004 Jul;30(7):476-81; discussion 475. doi: 10.1097/00004770-200407000-00005. PMID 15220641
- [Background] Siqueira JF Jr. Microbial causes of endodontic flare-ups. Int Endod J. 2003 Jul;36(7):453-63. doi: 10.1046/j.1365-2591.2003.00671.x. PMID 12823700
- [Background] Sathorn C, Parashos P, Messer H. Antibacterial efficacy of calcium hydroxide intracanal dressing: a systematic review and meta-analysis. Int Endod J. 2007 Jan;40(1):2-10. doi: 10.1111/j.1365-2591.2006.01197.x. PMID 17209826
- [Background] Caliskan MK. Nonsurgical retreatment of teeth with periapical lesions previously managed by either endodontic or surgical intervention. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Aug;100(2):242-8. doi: 10.1016/j.tripleo.2004.09.014. PMID 16037783
- [Background] Del Fabbro M, Taschieri S, Testori T, Francetti L, Weinstein RL. Surgical versus non-surgical endodontic re-treatment for periradicular lesions. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD005511. doi: 10.1002/14651858.CD005511.pub2. PMID 17636803
- [Background] Trope M. Relationship of intracanal medicaments to endodontic flare-ups. Endod Dent Traumatol. 1990 Oct;6(5):226-9. doi: 10.1111/j.1600-9657.1990.tb00423.x. PMID 2133314
- [Background] Gomes-Filho JE, Silva FO, Watanabe S, Cintra LT, Tendoro KV, Dalto LG, Pacanaro SV, Lodi CS, de Melo FF. Tissue reaction to silver nanoparticles dispersion as an alternative irrigating solution. J Endod. 2010 Oct;36(10):1698-702. doi: 10.1016/j.joen.2010.07.007. Epub 2010 Aug 24. PMID 20850681